CLINICAL TRIAL: NCT00003191
Title: A Phase I Study of Fenretinide (NSC #374551) in Children With High Risk Solid Tumors
Brief Title: Fenretinide in Treating Children With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02262; CCG-09709; CDR0000066023 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2003-11-26 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2006-08

CONDITIONS: Neuroblastoma; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: recurrent neuroblastoma; unspecified childhood solid tumor, protocol specific
MeSH Terms: conditions — Neuroblastoma | interventions — Fenretinide

ARMS (1):
- Arm I (Experimental): Patients receive oral fenretinide 3 times a day on days 1-7. Treatment repeats every 3 weeks for up to 8 courses. Patients may receive an additional 22 courses of therapy in the presence of stable or responding residual tumor. Patients with recurrent neuroblastoma, after prior myeloablative therapy with no measurable disease, will stop treatment after 8 courses. Cohorts of 3-6 patients receive escalating doses of fenretinide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity.
  Interventions: Drug: fenretinide

INTERVENTIONS:
Drug: fenretinide

SUMMARY:
Phase I trial to study the effectiveness of fenretinide in treating children who have solid tumors that have not responded to standard therapy. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of fenretinide (HPR) in children with high risk solid tumors.

II. Determine the toxicities of HPR in these patients. III. Determine the pharmacokinetics of HPR in these patients. IV. Determine the CSF level of HPR in patients whom cerebrospinal fluid is obtained for routine purposes while on this study.

V. Determine the effect of HPR on plasma retinol levels in these patients. VI. Determine the activity of HPR in these patients. VII. Determine the antitumor activity of HPR on minimal residual bone marrow disease in neuroblastoma.

OUTLINE: This is a dose escalation study.

Patients receive oral fenretinide 3 times a day on days 1-7. Treatment repeats every 3 weeks for up to 8 courses. Patients may receive an additional 22 courses of therapy in the presence of stable or responding residual tumor. Patients with recurrent neuroblastoma, after prior myeloablative therapy with no measurable disease, will stop treatment after 8 courses. Cohorts of 3-6 patients receive escalating doses of fenretinide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity.

Patients are followed until death.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant solid tumor that is refractory to conventional therapy or recurrent neuroblastoma treated with myeloablative therapy and autologous stem cell transplant in second complete or partial response
* Bone marrow metastases with granulocytopenia, anemia, and/or thrombocytopenia are eligible

PATIENT CHARACTERISTICS:

* Age: Under 21 at diagnosis
* Performance status: CCG 0-2
* Life expectancy: At least 2 months
* Absolute neutrophil count at least 750/mm3
* Platelet count at least 50,000/mm3
* Hemoglobin at least 7.0 g/dL
* Bilirubin no greater than 1.5 mg/dL
* SGOT and SGPT less than 2.5 times normal
* Creatinine no greater than 1.5 g/dL OR creatinine clearance at least 50 mL/min OR radioisotope GFR at least 50 mL/min
* Seizure disorders controlled with anticonvulsants allowed
* No CNS toxicity greater than grade 2
* Not pregnant
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* At least 1 month since prior autologous stem cell transplantation
* No prior allogeneic transplantation
* At least 2 weeks since prior chemotherapy (4 weeks for nitrosourea) and recovered
* No other concurrent chemotherapy
* No concurrent immunomodulating agents (including steroids)
* Concurrent corticosteroid therapy for increased intracranial pressure allowed
* Concurrent dexamethasone for CNS tumor allowed
* At least 2 weeks since prior radiotherapy
* Concurrent radiotherapy to localized lesions allowed
* At least 2 weeks since prior retinoids Prior isotretinoin or 9-cis-retinoic acid allowed

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 1998-03; Primary Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith G. Villablanca, MD, Study Chair — Children's Hospital Los Angeles
Locations (26):
- United States (25):
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia

REFERENCES:
- [Result] Children's Oncology Group (CCG 09709); Villablanca JG, Krailo MD, Ames MM, Reid JM, Reaman GH, Reynolds CP. Phase I trial of oral fenretinide in children with high-risk solid tumors: a report from the Children's Oncology Group (CCG 09709). J Clin Oncol. 2006 Jul 20;24(21):3423-30. doi: 10.1200/JCO.2005.03.9271. PMID 16849757
- [Result] Villablanca JG, Ames MW, Reid JM, et al.: Phase I trial of oral [N-(-4-hydroxyphenyl)retinamide] (4-HPR) in children with resistant/recurrent solid tumors: a children's cancer group study (CCG 09709). [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-1588, 2002.